CLINICAL TRIAL: NCT06845033
Title: Effects of Antagonizing the Ghrelin Receptor on Brain Food Cue Reactivity in Obesity
Acronym: LEAP2fMRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Anders Englund, Principal Investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-2306418; NNF23OC0084114 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEAP2 infusion (Active Comparator)
  Interventions: Other: LEAP2 infusion
- Placebo infusion (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: LEAP2 infusion — The LEAP2 infusion is a hormone infusion that is different from the placebo (saline) infusion
  Arms: LEAP2 infusion
Other: Placebo — Placebo infusion (saline) is different from the LEAP2 infusion
  Arms: Placebo infusion

SUMMARY:
The naturally occurring peptide hormone liver-expressed antimicrobial peptide 2 (LEAP2) in an antagonist/inverse agonist towards the ghrelin receptor. Ghrelin administration has previously been shown to increase food cue reactivity in brain regions related to appetite and reward using functional MRI scans.

The aim of this clinical study is to investigate the effects of LEAP2 infusion on food cue reactivity in brain regions related to appetite and reward. Since LEAP2 is an antagonist/inverse agonist towards the ghrelin receptor we hypothesize, that LEAP2 infusion will decrease food cue reactivity in the above-mentioned regions compared to placebo infusion.

Participants with obesity (BMI 30-50 kg/m2) will be included and complete two experimental days with either LEAP2 or placebo infusion in a randomized crossover manner. On experimental days, participants will undergo a MRI scan with functional and anatomical modalities.

The study will attribute to gain a deeper understanding of the ghrelin system and its interaction with appetite regulation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years at the time of inclusion
* Body mass index 30-50 kg/m2
* Men
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or present hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Glycated haemoglobin (HbA1c) ≥48 mmol/mol and/or type 2 diabetes requiring medical treatment
* Regular tobacco smoking or use of other nicotine-containing products
* Claustrophobia
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in food cue reactivity between experimental days | time 75 - 135 minutes
  The primary endpoint is the change in BOLD signals when viewing pictures of food vs. non-food. Differences will be compared between the two experimental days with infusion of placebo and LEAP2, respectively.

SECONDARY OUTCOMES:
Difference in appetite ratings | From baseline to end of infusion
  Difference in visual Analogue Scales (VASs) assessing appetite, satiety, and hunger sensations.
Changes in peptide hormone concentrations | From baseline to end of infusion
  Plasma/serum concentrations of LEAP2, growth hormone as well as other glucose- and appetite-regulating gut hormones

OTHER OUTCOMES:
Reactivity from Negative Emoition Reactivity Test (NERT) | time 75 - 135 minutes
  Change in BOLD signals when viewing pictures of that could cause stress (Negative Emoition Reactivity Test (NERT)). Differences will be compared between the two experimental days with infusion of placebo and LEAP2, respectively.
Plasma glucose | Through experimental day. From timepoints -15 to 135 min
  Change in plasma glucose concentration during the experimental days

IPD SHARING:
Plan to Share IPD: Undecided